CLINICAL TRIAL: NCT05378919
Title: Evaluation and Comparison of the Efficacy of a New Standard Pre-operative Chemotherapy for Stage II and III Colorectal Cancer According to the FOLFOX4 Regimen With Routine Chemoradiation Therapy
Brief Title: Neoadjuvant Therapy vs Standard Therapy in Locally Advanced Rectal Cancer
Acronym: RECTUM2015
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Rita Ambraziene, Sub-Investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECTUM2015
Record Dates: First submitted 2022-05-08; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Neoadjuvant Therapy in Rectal Cancer, Radiotherapy, FOLFOX
MeSH Terms: interventions — Fluorouracil; Folic Acid; Drug Therapy; Clinical Protocols; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Control): Radiotherapy + fluorouracil (Active Comparator): Chemoradiotherapy 5 weeks (50 Grays (Gy), 2 Gy/session; 25 fractions) + fluorouracil/leucovorin 400 mg/m² 1-4 day the first and fifth weeks of radiotherapy) , then 6-8 weeks after chemoradiation, surgery, followed by adjuvant chemotherapy for 4-6 months, either Folfox4 or fluorouracil, depending on the center's choice.
  Interventions: Radiation: Radiotherapy 50 Gy; Drug: Fluorouracil/folic acid
- Arm B (Experimental): Chemotherapy with Oxaliplatin, fluorouracil, folinic acid (FOLFOX4) regimen (Experimental): Neoadjuvant CT FOLFOX4, 8 cycles (ca. 4 months; each cycle = 2 weeks):
  oxaliplatin: 85 mg/m² in 2 hours at D1; folinic acid: 100 mg/m² simultaneously in 2 hours at D1 and D2 during the Oxaliplatin; bolus 5-fluorouracil (5-FU) 400mg/m² D1+D2; infusion 5-fluorouracil (5-FU): 600 mg/m² continuous infusion during 22hours at D1 and D2, every 14 days during 42 months (8 cycles).
  Interventions: Drug: Chemotherapy in regimen with Oxaliplatin, fluorouracil, folinic acid (FOLFOX4); Radiation: Radiotherapy 50 Gy

INTERVENTIONS:
Radiation: Radiotherapy 50 Gy — Radiotherapy 50 Gy 5 radiations per week of 2 Gy for 5 weeks
  Arms: Arm A (Control): Radiotherapy + fluorouracil
Drug: Fluorouracil/folic acid — Fluorouracil 400 mg/m² D1-4 and folic acid 20mg/m2 D1-4 the first and fifth weeks of radiotherapy
  Arms: Arm A (Control): Radiotherapy + fluorouracil
Drug: Chemotherapy in regimen with Oxaliplatin, fluorouracil, folinic acid (FOLFOX4) — oxaliplatin: 85 mg/m² in 2 hours at D1; folinic acid: 100 mg/m² simultaneously in 2 hours at D1 and D2 during the Oxaliplatin; bolus 5-fluorouracil (5-FU) 400mg/m² D1+D2; infusion 5-fluorouracil (5-FU): 600 mg/m² continuous infusion during 22hours at D1 and D2, every 14 days during 42 months (8 cycles).
  Arms: Arm B (Experimental): Chemotherapy with Oxaliplatin, fluorouracil, folinic acid (FOLFOX4) regimen
Radiation: Radiotherapy 50 Gy — Chemoradiotherapy 5 weeks (50 Grays (Gy), 2 Gy/session; 25 fractions) + fluorouracil/leucovorin 400 mg/m² 1-4 day the first and fifth weeks of radiotherapy.
  FOLOFX4 will be administrated for 8 cycles over a 16 week period. Patients will undergo re-staging within 6 weeks of their 8th cycle of FOLFOX. This will include MRI of the pelvis. If the reassessment reveals that there has been no disease progression compared to the pre-treatment evaluation and the patient remains a candidate for an R0 resection, the patient will proceed to definitive rectal cancer surgery within 8 weeks from the last chemotherapy dose. If the surgical oncologist's reassessment reveals that the patient is not a candidate for an R0 resection, the patient will proceed to standard pre-operative radiation with synchronous fluorouracil.
  Arms: Arm B (Experimental): Chemotherapy with Oxaliplatin, fluorouracil, folinic acid (FOLFOX4) regimen

SUMMARY:
Phase II, Multicenter, Open-label, Randomized Study evaluating neoadjuvant chemotherapy (FOLFOX4) in patients with stage II and III colorectal cancer with standard chemoradiation Defined by Magnetic Resonance Imaging

DETAILED DESCRIPTION:
This is a biomedical research, phase II, multicenter, open-label, randomized study, comparing neoadjuvant CT with FOLFOX4, versus immediate preoperative chemoradiotherapy (CRT), in patients with locally advanced rectal cancer. Randomization in a 1: 1 ratio, neoadjuvant chemotherapy or chemoradiation. The purpose of the study is to evaluate the efficacy, tolerability, and comparability of new standard preoperative chemotherapy with FOLFOX4 in patients with stage II and III colorectal cancer compared to routine chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with rectal adenocarcinoma;
* radiologically measurable tumor size;
* general condition (ECOG 0-2 points);
* stage II or III rectal tumor clinically (pelvic MRI and endorectal ultrasound),
* in the absence of long-term spread of the disease (confirmed by radiological examinations (computed tomography of the thorax and abdomen));
* during preoperative proctoscopy, the tumor is detected 0 -15 cm from the anus;
* Blood tests 28 days before the start of treatment:

and general blood count: neutrophils greater than 1.5x10 9 / l, platelets greater than 100 x 10 9 / l, Hemoglobin greater than 80 g / l, liver enzymes (Aspartate aminotransferase (AST/GOT), alanine aminotransferase (ALT/GPT) not more than 3 times upper limit), and renal function (creatinine up to 1.5 times the upper limit of normal) is normal; women of childbearing potential - negative pregnancy test;

• A signed informed consent form.

Exclusion Criteria:

* patients with signs of intestinal obstruction at the start of treatment;
* previous lower abdominal radiation therapy;
* other tumors over a five-year period;
* pregnant or breastfeeding women;
* men and women of childbearing potential who do not agree to use adequate contraception;
* Patient co-morbidities that would make the patient unsuitable for this study or significantly interfere with the assessment of safety and toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 year
  To compare the 3-year disease-free survival between the investigational arm and the control arm.

SECONDARY OUTCOMES:
Overall survival | 7 year
  Overall survival will be defined as the time from randomisation to the time of occurrence of the first death regardless to its cause. Patients alive at the time of analysis will be censored at the date of the last follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Rita Ambraziene, Kaunas, Lithuania